CLINICAL TRIAL: NCT02943057
Title: Intra-cameral Penetration and Efficacy of Ganciclovir Following Topical Administration of 2% Ganciclovir Eye Drop for CMV Anterior Uveitis / Endotheliitis
Brief Title: Topical 2% Ganciclovir Eye Drop for CMV Anterior Uveitis / Endotheliitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Soon Phaik Chee, Senior Consultant & HOD, Singapore National Eye Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1226/32/2015
Record Dates: First submitted 2016-10-18; First posted 2016-10-24 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2024-04

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2% guttae Ganciclovir (Experimental): 2% guttae Ganciclovir 5 times a day for 6 weeks
  Interventions: Drug: 2% guttae ganciclovir

INTERVENTIONS:
Drug: 2% guttae ganciclovir — 2% guttae ganciclovir 5 times a day for 6 weeks

SUMMARY:
25 patients who are diagnosed with Cytomegalovirus (CMV) anterior segment infection, either uveitis or endotheliitis, will be started on 2% guttae ganciclovir, 1 drop 5 times a day for 6 weeks.

Following 6 weeks of continuous application of 2% guttae ganciclovir, patient will be reviewed at the clinic within 3 hours following the last application of topical ganciclovir and clinical features will be documented for activity assessment. An aqueous sample 0.2ml is drawn. 0.1ml will be sent for RT-PCR for CMV viral load and another 0.1ml will be sent for ganciclovir drug level by HPLC method.

DETAILED DESCRIPTION:
This is non-randomised single armed prospective, cross-sectional, interventional clinical study.

25 patients who are diagnosed with Cytomegalovirus (CMV) anterior segment infection, either uveitis or endotheliitis, at the investigators clinic in Singapore National Eye Centre, who have a positive aqueous real time PCR (RT-PCR) and/or positive tetraplex PCR for CMV and have not had any form of ganciclovir treatment in the past 1 month, will be recruited in the study after taking an informed consent. This will also include the patients who have never been treated with antiviral therapy and those with recurrent disease and have not had any form of ganciclovir treatment for past 1 month.

The clinical features of the active disease will be recorded in the data collection sheet and will include, documentation of the state of the cornea, KPs, AC cells, flare, flare meter reading (where possible), central corneal thickness, Intra ocular pressure (IOP) and C:D ratio.

All patients will be started on 2% guttae ganciclovir, 1 drop 5 times a day.

2% Guttae ganciclovir will be prepared from vials of ganciclovir powder for ganciclovir intravenous infusion using aseptic method.

Following 6 weeks of continuous application of 2% guttae ganciclovir, patient will be reviewed at the clinic within 3 hours following the last application of topical ganciclovir.

1. Clinical features mentioned above will be documented for activity assessment
2. Following irrigation of the conjunctival sac with 100ml of N/S to wash out any residual drug, aseptic technique is practised before an aqueous sample 0.2ml is drawn. 0.1ml will be sent for RT-PCR for CMV viral load and another 0.1ml will be sent for ganciclovir drug level by HPLC method.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and above
* Patients who are diagnosed with anterior uveitis or endotheliitis with a positive aqueous real time PCR (RT-PCR) and/or positive tetraplex PCR for Cytomegalovirus (CMV)
* Patients with relapses and recurrent anterior segment disease that is PCR positive for CMV in aqueous
* Have not been on any form of (topical, local or systemic) ganciclovir therapy for the past 1 month
* Consent to undergo anterior chamber tap and give aqueous and tear samples for the study
* Able to undergo relevant tests (e.g. laser flare cell photometry)
* Able to come for subsequent follow-up visits
* Ability to provide informed consent

Exclusion Criteria:

* CMV anterior uveitis with associated retinitis
* Other causes of hypertensive anterior uveitis / endotheliitis such as HSV, VZV infection
* Patients who have been on any form of (topical, local or systemic) ganciclovir therapy for the past1 month.
* Patients who are allergic to ganciclovir
* Patients who will require systemic or intra-vitreal ganciclovir therapy
* Immunocompromised patients
* Positive for HIV, Hep B and Hep C
* Not keen on participating in the study
* Patients who are incapable, either by law or mental state, of giving consents in their own right.
* Patients who are either unable or unwilling to keep scheduled appointments and adhere to the other aspects of the protocol
* Patients who are pregnant or breastfeeding
* Any other specified reason as determined by the clinical investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2024-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Median concentration of ganciclovir in aqueous by HPLC-Mass spectrometry end of week 6 | 6 weeks
  Ganciclovir concentration in aqueous will be measured by HPLC-Mass spectrometry at the end of week 6

SECONDARY OUTCOMES:
Clinical efficacy in clearing CMV viral load and resolution of anterior uveitis/endotheliitis following 6 weeks of treatment | 6 weeks
  Clinical efficacy will be measured by resolution of anterior uveitis/ endotheliitis and aqueous tap negative for CMV realtime PCR at the end of week 6

CONTACTS AND LOCATIONS:
Overall Officials: SP Chee, Study Chair — Singapre national eye centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No